CLINICAL TRIAL: NCT01178320
Title: Carotid Plaque Characteristics by MRI in AIM-HIGH
Brief Title: Carotid Plaque Characteristics by MRI in AIM-HIGH (Carotid MRI Substudy)
Status: Completed | Type: Observational
Sponsor: University of Washington (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Xue-Qiao Zhao, Professor, University of Washington
Other Study IDs: 627; R01HL088214 (NIH)
Record Dates: First submitted 2010-08-05; First posted 2010-08-10 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Coronary Artery Disease; Carotid Artery Diseases; Atherosclerosis
Keywords: Magnetic Resonance Imaging; Atherosclerotic Plaque; Lipid Lowering Therapy
MeSH Terms: conditions — Coronary Artery Disease; Carotid Artery Diseases; Atherosclerosis; Plaque, Atherosclerotic | interventions — Simvastatin; Niacin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Simvastatin: Participants in the main AIM-HIGH study who are receiving simvastatin.
  Interventions: Drug: Simvastatin, simvastatin plus extended-release niacin
- Simvastatin and Extended-Release Niacin: Participants in the main AIM-HIGH study who are receiving simvastatin and extended-release niacin.
  Interventions: Drug: Simvastatin, simvastatin plus extended-release niacin

INTERVENTIONS:
Drug: Simvastatin, simvastatin plus extended-release niacin — Participants will be enrolled in this substudy only if they are candidates for the main AIM-HIGH study (NCT00120289). Participants will be randomly assigned to simvastatin or simvastatin plus niacin as a part of the main AIM-HIGH protocol, and adjustments in simvastatin and/or niacin doses will be made as per the protocol for the main AIM-HIGH study.
  Other Names: simvastatin; Zocor; niacin; Niaspan

SUMMARY:
Heart attacks and strokes caused by the unstable atherosclerotic plaques remain the leading cause of death in the United States. Unstable plaques often have more fat than stable plaques. This study will investigate if a treatment with LDL-lowering plus HDL-raising compared with LDL-lowering alone would more effectively reduce the plaque fat content assessed by magnetic resonance imaging (MRI), therefore, further reducing heart attacks and strokes.

DETAILED DESCRIPTION:
Although studies have suggested that plaque morphology and composition are important determinants of plaque stability, our understanding on plaque tissue components is mainly from histological studies until recent development in MRI technique. A low level of HDL is associated with higher risk of cardiovascular events and increased amount of lipid content in the carotid plaques. Treatment with LDL-lowering plus HDL-raising compared with LDL-lowering alone more effectively protects against atherosclerosis progression. It is widely believed that HDL or its apolipoproteins mediate the removal of excess free cholesterol from peripheral cells and the cholesterol is delivered via either LDL or HDL to the liver for excretion into the bile. However, it has not been tested and approved in human atherosclerotic condition in vivo. The NIH/Abbott-funded multi-center AIM-HIGH trial is designed to compare the clinical efficacy of LDL-lowering alone with statin versus LDL-lowering plus HDL-raising with statin plus nicotinic acid combination therapy in patients with established vascular disease and high triglycerides and low HDL.

We propose to conduct a carotid MRI sub-study in 220 subjects enrolled in AIM-HIGH to investigate the important vascular biological mechanisms of HDL-raising therapy. Image collection will occur at 3 timepoints. The hypotheses and specific aims are:

* (1) To test the primary hypothesis that compared with LDL-lowering alone, intensive LDL-lowering plus HDL-raising therapy decreases the mean plaque lipid composition in carotid arteries assessed by MRI.
* (2) To test the hypothesis that compared with LDL-lowering alone, intensive LDL-lowering plus HDL-raising therapy decreases the plaque burden including volume and wall thickness.
* (3) To test the hypothesis that increased plaque lipid composition or vessel wall thickness by MRI is associated with increased risk of cardiovascular events.
* (4)To test a hypothesis that LDL-lowering plus HDL-raising, compared to LDL-lowering alone, will promote more rapid plaque lipid depletion. And determine the time-course of atherosclerotic plaque lipid depletion during lipid therapy.
* (5) To examine the association of clinical risk factors, lipids, lipoprotein heterogeneity, inflammatory markers and carotid plaque characteristics.

This MRI sub-study offers a unique opportunity to investigate the effectiveness of LDL-lowering plus HDL-raising therapy on human atherosclerotic plaque in vivo, to examine the association of plaque characteristics both lipid composition and volume assessed by MRI and cardiovascular outcome, and to gain novel insights in our understanding of atherosclerotic plaque pathology and the mechanisms of intensive lipid management in preventing cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Eligible for main AIM-HIGH study (NCT00120289)
* Medically able to undergo MRI procedure
* Willing to provide informed consent for participation in this substudy

Exclusion Criteria:

* Uses pacemaker or has metallic implants
* History of bilateral carotid endarterectomy
* Glomerular filtration rate less than 60 mL/min/1.73 m^2

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the main AIM-HIGH study (NCT00120289)
Sampling Method: Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2008-03; Primary Completion 2013-04 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Mean plaque lipid composition in carotid arteries assessed by MR | Through 24Months post AIM-HIGH Randomization
  To test the primary hypothesis that compared with LDL-lowering alone, intensive LDL-lowering plus HDL-raising therapy decreases the mean plaque lipid composition in carotid arteries assessed by MRI.

SECONDARY OUTCOMES:
Additional plaque characteristics as assessed by MRI | Through 24Months post AIM-HIGH Randomization
  To test the additional hypotheses regarding plaque burden, plaque lipid depletion time course, association with cardiovascular event risk and lipid characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Xue-Qiao Zhao, MD, Principal Investigator — University of Washington
Locations (19):
- United States (15):
  - Cardiovascular Consultants, Phoenix, Arizona
  - Long Beach VA Medical Center, Long Beach, California
  - University of Southern California, Los Angeles, California
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Philadelphia VA Medical Center, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Kelsey Research Foundation, Houston, Texas
  - Methodist Hospital, Houston, Texas
  - Harborview Medical Center, Seattle, Washington
  - University of Washington, Seattle, Washington
  - Puget Sound VA Medical Center, Seattle Campus, Seattle, Washington
- Canada (4):
  - Heart Health Institute, Calgary, Alberta
  - University of Calgary, Calgary, Alberta
  - Vancouver General Hospital, Vancouver, British Columbia
  - University of Western Ontario, London, Ontario

REFERENCES:
- [Result] Hippe DS, Phan BAP, Sun J, Isquith DA, O'Brien KD, Crouse JR, Anderson T, Huston J, Marcovina SM, Hatsukami TS, Yuan C, Zhao XQ. Lp(a) (Lipoprotein(a)) Levels Predict Progression of Carotid Atherosclerosis in Subjects With Atherosclerotic Cardiovascular Disease on Intensive Lipid Therapy: An Analysis of the AIM-HIGH (Atherothrombosis Intervention in Metabolic Syndrome With Low HDL/High Triglycerides: Impact on Global Health Outcomes) Carotid Magnetic Resonance Imaging Substudy-Brief Report. Arterioscler Thromb Vasc Biol. 2018 Mar;38(3):673-678. doi: 10.1161/ATVBAHA.117.310368. Epub 2018 Jan 4. PMID 29301785
- [Result] Sun J, Zhao XQ, Balu N, Hippe DS, Hatsukami TS, Isquith DA, Yamada K, Neradilek MB, Canton G, Xue Y, Fleg JL, Desvigne-Nickens P, Klimas MT, Padley RJ, Vassileva MT, Wyman BT, Yuan C. Carotid magnetic resonance imaging for monitoring atherosclerotic plaque progression: a multicenter reproducibility study. Int J Cardiovasc Imaging. 2015 Jan;31(1):95-103. doi: 10.1007/s10554-014-0532-7. Epub 2014 Sep 13. PMID 25216871
- [Result] Chen H, Sun J, Kerwin WS, Balu N, Neradilek MB, Hippe DS, Isquith D, Xue Y, Yamada K, Peck S, Yuan C, O'Brien KD, Zhao XQ. Scan-rescan reproducibility of quantitative assessment of inflammatory carotid atherosclerotic plaque using dynamic contrast-enhanced 3T CMR in a multi-center study. J Cardiovasc Magn Reson. 2014 Aug 1;16(1):51. doi: 10.1186/s12968-014-0051-7. PMID 25084698
- [Result] Zhao XQ, Hatsukami TS, Hippe DS, Sun J, Balu N, Isquith DA, Crouse JR 3rd, Anderson T, Huston J 3rd, Polissar N, O'Brien K, Yuan C; AIM-HIGH Carotid MRI Sub-study Investigators. Clinical factors associated with high-risk carotid plaque features as assessed by magnetic resonance imaging in patients with established vascular disease (from the AIM-HIGH Study). Am J Cardiol. 2014 Nov 1;114(9):1412-9. doi: 10.1016/j.amjcard.2014.08.001. Epub 2014 Aug 13. PMID 25245415
- [Derived] Zhao XQ, Sun J, Hippe DS, Isquith DA, Canton G, Yamada K, Balu N, Crouse JR 3rd, Anderson TJ, Huston J 3rd, O'Brien KD, Hatsukami TS, Yuan C; AIM-HIGH Carotid MRI Substudy Investigators. Magnetic Resonance Imaging of Intraplaque Hemorrhage and Plaque Lipid Content With Continued Lipid-Lowering Therapy: Results of a Magnetic Resonance Imaging Substudy in AIM-HIGH. Circ Cardiovasc Imaging. 2022 Nov;15(11):e014229. doi: 10.1161/CIRCIMAGING.122.014229. Epub 2022 Nov 15. PMID 36378778
- [Derived] O'Brien KD, Hippe DS, Chen H, Neradilek MB, Probstfield JL, Peck S, Isquith DA, Canton G, Yuan C, Polissar NL, Zhao XQ, Kerwin WS. Longer duration of statin therapy is associated with decreased carotid plaque vascularity by magnetic resonance imaging. Atherosclerosis. 2016 Feb;245:74-81. doi: 10.1016/j.atherosclerosis.2015.11.032. Epub 2015 Dec 1. PMID 26708287